CLINICAL TRIAL: NCT01581125
Title: Sleep Duration Required to Restore Performance During Chronic Sleep Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth B. Klerman, Associate Professor, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NIH R01 HL114088-01
Record Dates: First submitted 2012-03-22; First posted 2012-04-19 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Sleep; Sleep Deprivation; Insufficient Sleep Syndrome
Keywords: Inpatients; Health Normalcy; circadian rhythm
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep:wake 2 (Experimental): Sleep and wake durations for arm 2 for inpatient portion of protocol. .There are a variety of sleep and wake durations during the protocol; some of these are longer and some are shorter and some are the same as in arm 1.
  Interventions: Behavioral: Sleep:wake 2
- Sleep:wake 1 (Experimental): Sleep and wake durations for arm 1 of the inpatient portion of the protocol. There are a variety of sleep and wake durations during the protocol; some of these are longer and some are shorter and some are the same as in arm 2.
  Interventions: Behavioral: Sleep:wake 1

INTERVENTIONS:
Behavioral: Sleep:wake 1 — Sleep and Wake durations for arm 1
  Arms: Sleep:wake 1
Behavioral: Sleep:wake 2 — Sleep and Wake durations for arm2
  Arms: Sleep:wake 2

SUMMARY:
The purpose of this study is to test the hypothesis that sleep and performance depend on length of time awake, length of time asleep, the amount of sleep over several sleep episodes, and circadian phase.

DETAILED DESCRIPTION:
The purpose of this study is to test the hypothesis that sleep and performance depend on length of time awake, length of time asleep, the amount of sleep over several sleep episodes, and circadian phase. Inpatient sleep and performance data will be collected from healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Prescription medications

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2012-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Psychomotor Vigilance Task (PVT) performance | PVT during waking for arms 1 and 2 during the 32-day inpatient portion of the protocol
  PVT metrics are reaction time. It is measured when the participants are awake during the inpatient portion of the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth B Klerman, MD PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] McHill AW, Hull JT, Cohen DA, Wang W, Czeisler CA, Klerman EB. Chronic sleep restriction greatly magnifies performance decrements immediately after awakening. Sleep. 2019 May 1;42(5):zsz032. doi: 10.1093/sleep/zsz032. PMID 30722039
- [Derived] McHill AW, Hull JT, McMullan CJ, Klerman EB. Chronic Insufficient Sleep Has a Limited Impact on Circadian Rhythmicity of Subjective Hunger and Awakening Fasted Metabolic Hormones. Front Endocrinol (Lausanne). 2018 Jun 12;9:319. doi: 10.3389/fendo.2018.00319. eCollection 2018. PMID 29946297